CLINICAL TRIAL: NCT04617691
Title: An Open-label, Randomized, Parallel-group Study to Assess the Bioequivalence of the Intravenous Formulation of Guselkumab Using Prefilled Syringes Assembled in an UltraSafe Plus Passive Needle Guard and Intravenous Formulation of Guselkumab Using Final Vialed Product in Healthy Participants
Brief Title: A Study of Intravenous Formulation of Guselkumab Using Prefilled Syringes and Final Vialed Product in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108895; CNTO1959EDI1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-11-03; First posted 2020-11-05 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: Tremfya
MeSH Terms: interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Guselkumab PFS-U (Experimental): Participants will receive single intravenous (IV) guselkumab formulation using UltraSafe Plus Passive Needle Guards (PFS-U) to create the IV solution.
  Interventions: Drug: Guselkumab
- Group 2: Guselkumab FVP (Experimental): Participants will receive single IV guselkumab formulation using Final Vialed Product (FVP) to create the IV solution.
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered as IV solution derived from FVP or PFS-U.

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of an intravenous (IV) administration of the guselkumab formulation using UltraSafe Plus Passive Needle Guard (PFS-U) to create the IV solution versus the guselkumab formulation using Final Vialed Product (FVP) (IV) to create the IV solution.

ELIGIBILITY:
Inclusion Criteria:

* Be healthy on the basis of physical examination, medical history, vital signs and electrocardiogram (ECG) performed at screening. Any abnormalities must be considered not clinically significant and this determination must be recorded in the participant's source documents and initialed by the investigator
* Be healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* A female participant must have a negative pregnancy test result at screening and baseline (Day -1) and while enrolled in this study
* Must be a non-user or light user of tobacco products (not smoke more than 10 cigarettes or equivalent a day for at least 6 months prior to screening), including all nicotine use, example, cigarettes (including e-cigarettes or the equivalent of e-cigarettes), cigars, chewing tobacco, patch, gum
* Participant is considered eligible according to the following tuberculosis (TB) screening criteria: (a) have no history of latent or active TB before screening; (b) have no signs or symptoms suggestive of active TB upon medical history and/or physical examination; (c) have had no recent close contact with a person with active TB; (d) have a negative QuantiFERON-TB test result within 28 days prior to the administration of study intervention

Exclusion Criteria:

* History of any clinically significant medical illness or medical disorders the investigator considers should exclude the participant, including (but not limited to), neuromuscular, hematological disease, immune deficiency state, respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease
* History of malignancy before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Has a current chronic infection, prior history of recurrent infection, or an active infection
* Received any systemic immunosuppressant agent (other than a short course of corticosteroids for minor inflammatory conditions) within 6 months before and during screening and administration of study intervention
* Has a positive urine drug or alcohol screen during screening or at admission (Day -1)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) | Up to Day 85
  Cmax is defined as maximum observed serum concentration.
Area Under The Serum Concentration Versus Time Curve From Time 0 to Infinity Based on Extrapolation of The Terminal Phase (AUC[0-infinity]) | Up to Day 85
  AUC(0-infinity) is defined as area under the serum concentration vs time curve from time 0 to infinity based on extrapolation of the terminal phase.

SECONDARY OUTCOMES:
Percentage of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to Day 85
  An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Percentage of Participants with Serious Adverse Events (SAEs) | Up to Day 85
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Percentage of Participants with Clinically Significant Changes in Vital Signs | Up to Day 85
  Percentage of participants with clinically significant changes in vital signs (including temperature (oral), pulse/heart rate, respiratory rate, and blood pressure) will be reported.
Percentage of Participants with Clinically Significant Changes in Physical Examinations | Up to Day 85
  Percentage of participants with clinically significant changes in physical examinations (including general appearance, respiratory, cardiovascular, assessment of the skin at or around the intravenous [IV] administration area) will be reported.
Percentage of Participants with Clinically Significant Changes in Laboratory Safety Tests | Up to Day 85
  Percentage of participants with clinically significant changes in laboratory safety tests (such as serum chemistry, hematology and urinalysis) will be reported.
Percentage of Participants with Antibodies to Guselkumab | Up to Day 85
  Percentage of participants with antibodies to guselkumab will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency